CLINICAL TRIAL: NCT02268331
Title: Comparison of Active vs. Passive Surveillance to Collect Adverse Events After Chiropractic Manual Therapy in the Children
Brief Title: Comparison of Active vs. Passive Surveillance to Collect Adverse Events
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Surveillance
Record Dates: First submitted 2014-10-10; First posted 2014-10-20 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2016-09

CONDITIONS: Adverse Events
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Surveillance (Experimental): For 60 consecutive pediatric visits, patients will be asked to complete a PRE & POST form to capture adverse events (AEs) that occur up to 1 week after treatment. The PRE-treatment form will be completed prior to the start of the visit. The POST-treatment form will be completed after the treatment visit and mailed directly to the investigative team.
  The providers will collect data on the treatment provided on the same 60 pediatric patients. The treatment provided is at the discretion of the doctors. If a moderate, serious, or severe AE occurs, the provider will complete the AE form with detailed information about potential risk factors and patient outcomes.
  Interventions: Other: Active Surveillance
- Passive Surveillance (Active Comparator): All doctors allocated to this arm will be provided with a username and password with an established chiropractic passive surveillance reporting and learning online system (CPiRLS) in the UK. If a patient safety incident occurs in their office or an adverse event (AE), the provider will complete a report on the CPiRLS website. The providers can record events that occur during the time period of 60 pediatric visits.
  Treatment provided during these treatments is at the doctor's discretion.
  Interventions: Other: Passive Surveillance

INTERVENTIONS:
Other: Active Surveillance
  Arms: Active Surveillance
Other: Passive Surveillance
  Arms: Passive Surveillance

SUMMARY:
This cluster randomized trial will be the first to specifically evaluate passive versus active surveillance methods collection of adverse events (AEs). The evaluation of these methods will be performed within the chiropractic healthcare profession, specifically among those who treat children. To date there is no mandatory reporting and learning as part of their profession. In Europe, a passive (voluntary) reporting and learning online system (CPiRLS) has been created and will be utilized in this study for the passive reporting and learning arm.

Manual therapy is the most common intervention provided by the chiropractic profession and is the most commonly sought provider-administrated complementary and alternative therapy in the United States pediatric population. This study will randomize participating doctors of chiropractic who often treat children, to of one of two arms (active vs. passive reporting and learning) to evaluate the quantity and quality of AE data collected.

ELIGIBILITY:
Inclusion Criteria:

* Licensed doctors of chiropractic who provide manual therapy in US or Canada
* Willing to collect data per protocol for 60 consecutive pediatric (13 years of age and younger) patients

Exclusion Criteria:

- Doctors of chiropractic and patient participation will be limited to those that speak / read English.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Adverse event occurring after treatment | Up to one week after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sunita Vohra, MD, FRCPC, MSc, Principal Investigator — University of Alberta
Locations (1):
- CARE, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Pohlman KA, Carroll L, Tsuyuki RT, Hartling L, Vohra S. Active versus passive adverse event reporting after pediatric chiropractic manual therapy: study protocol for a cluster randomized controlled trial. Trials. 2017 Dec 1;18(1):575. doi: 10.1186/s13063-017-2301-0. PMID 29191232